CLINICAL TRIAL: NCT01520987
Title: Randomized, Double-Blinded, Placebo-Controlled, Multiple Ascending Dose Study to Compare the Pharmacokinetics of BIA 9-1067 in Healthy Japanese and Caucasian Subjects
Brief Title: Pharmacokinetics of BIA 9-1067 in Healthy Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-91067-126
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Results first posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; BIA 9-1067
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Caucasian 5 mg OPC (Experimental): OPC, opicapone, BIA 9-1067
  Interventions: Drug: BIA 9-1067
- Caucasian 25 mg OPC (Experimental): OPC, opicapone, BIA 9-1067
  Interventions: Drug: BIA 9-1067
- Caucasian 50 mg OPC (Experimental): OPC, opicapone, BIA 9-1067
  Interventions: Drug: BIA 9-1067
- Caucasian Placebo (Placebo Comparator): Placebo, PLC
  Interventions: Drug: Placebo
- Japanese 5 mg OPC (Experimental): OPC, opicapone, BIA 9-1067
  Interventions: Drug: BIA 9-1067
- Japanese 25 mg OPC (Experimental): OPC, opicapone, BIA 9-1067
  Interventions: Drug: BIA 9-1067
- Japanese 50 mg OPC (Experimental): OPC, opicapone, BIA 9-1067
  Interventions: Drug: BIA 9-1067
- Japanese Placebo (Placebo Comparator): Placebo, PLC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIA 9-1067 — 5 mg, 25 mg, and 50 mg of BIA 9-1067 (once-daily).
  Arms: Caucasian 25 mg OPC; Caucasian 5 mg OPC; Caucasian 50 mg OPC; Japanese 25 mg OPC; Japanese 5 mg OPC; Japanese 50 mg OPC
Drug: Placebo — once-daily
  Arms: Caucasian Placebo; Japanese Placebo

SUMMARY:
To assess the pharmacokinetics of BIA 9-1067 in healthy Japanese subjects

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled, multiple ascending dose, parallel-group, pharmacokinetic (PK) and pharmacodynamic (PD) study

ELIGIBILITY:
Inclusion Criteria:

* Men or nonlactating and nonpregnant women;
* Caucasian or Japanese subjects. Caucasian subjects are subjects of European descent; Japanese subjects must be first or second generation. Generations will be defined as follows:

  1. First generation Japanese are subjects who may be living outside Japan but were born in Japan to parents of Japanese descent.
  2. Second generation Japanese are subjects who were born outside of Japan to first generation Japanese parents.
* Aged 18 to 65 years;
* Body weight ≥50 kg;
* Within BMI range 18.5 to 30 kg/m2, inclusive;
* Healthy, as determined by the Investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead ECG. Creatinine and ALT levels must be strictly within the normal range for eligibility at Check-in;
* Women of nonchildbearing potential must be surgically sterile (hysterectomy, oophorectomy, or tubal ligation) or postmenopausal for ≥1 year;
* Women of childbearing potential must be using an effective nonhormonal method of contraception (intrauterine device or intrauterine system; condom or occlusive cap [diaphragm or cervical or vault caps] with spermicidal foam or gel or film or cream or suppository; true abstinence; or vasectomized male partner, provided that he is the sole partner of that subject) for a period of at least 1 month before and after dose administration. Women of childbearing potential must have a negative pregnancy test result within 48 hours before the start of the first investigational medicinal product (IMP) administration. Hormonal contraceptives will not be allowed because the effect of BIA 9 1067 on the metabolism of hormonal contraceptives and vice versa is not yet known;
* Nonsmokers, defined as having smoked ≤10 cigarettes per week for the 3 months prior to dosing, abstained from smoking for 7 days prior to Check-in, and having a negative cotinine level ≤500 ng/mL at Check-in;
* Have a high probability for compliance with and completion of the study, in the opinion of the Investigator;
* Able to comprehend and willing to sign an ICF.

Exclusion Criteria:

* Presence or history of any disorder that may prevent the successful completion of the study;
* History of multiple and/or severe allergies to drugs or foods or a history of anaphylactic reactions;
* Known or suspected allergy or other adverse drug reactions to the trial product or related products (eg, tolcapone or entacapone);
* History of alcoholism or excessive daily alcohol consumption within the past year. Excessive alcohol consumption is regarded as an average weekly intake of more than 14 units for women and 21 units for men (1 unit of alcohol = 8 to 10 g and is approximately equivalent to 1 glass of wine or 250 mL of beer or a standard measure of spirits);
* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease, as judged by the Investigator or Sponsor's Medical Monitor;
* Any clinically important deviation from normal limits in physical examination, vital signs, or 12-lead ECGs, as judged by the Investigator or Sponsor's Medical Monitor;
* Acute disease state (eg, nausea, vomiting, fever, diarrhea) within 7 days of Study Day 1;
* Positive serologic findings for HIV antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus antibodies (anti-HCV);
* Positive screen for drugs of abuse and alcohol;
* Recent history or presence of any disorder that may interfere with the absorption, distribution, metabolism, or excretion of BIA 9 1067;
* Positive pregnancy test result for WOCBP only;
* Consumption of any caffeine-containing products (eg, coffee, tea, chocolate, or cola), grapefruit, grapefruit-containing products, or alcoholic beverages from 48 hours before Study Day 1 until Discharge (Day 16);
* Involvement in other investigational studies of any type within 30 days of BIA 9-1067 administration;
* Donation of blood within 90 days of Study Day 1;
* Use of any prescription drug within 30 days of IMP administration unless deemed acceptable by the Principal Investigator (PI) and Medical Monitor;
* Use of any over-the-counter drugs including herbal supplements (except for the occasional use of acetaminophen and vitamins ≤100% recommended daily allowance) within 14 days of Study Day 1 unless deemed acceptable by the PI and Medical Monitor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haejung Marr, MD, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit, Inc., Honolulu, Hawaii, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Caucasian 5 mg OPC; Caucasian 25 mg OPC; Caucasian 50 mg OPC; Japanese 5 mg OPC; Japanese 25 mg OPC; Japanese 50 mg OPC: OPC, opicapone, BIA 9-1067 (once-daily).
Period: Overall Study
Arm/Group | Caucasian 5 mg OPC | Caucasian 25 mg OPC | Caucasian 50 mg OPC | Caucasian Placebo | Japanese 5 mg OPC | Japanese 25 mg OPC | Japanese 50 mg OPC | Japanese Placebo
Started | 13 | 12 | 11 | 15 | 14 | 14 | 12 | 14
Dosed | 13 | 12 | 11 | 15 | 14 | 14 | 12 | 14
Completed | 12 | 12 | 11 | 15 | 14 | 13 | 12 | 14
Not Completed | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caucasian 5 mg OPC | Caucasian 25 mg OPC | Caucasian 50 mg OPC | Caucasian Placebo | Japanese 5 mg OPC | Japanese 25 mg OPC | Japanese 50 mg OPC | Japanese Placebo | Total
Number analyzed (Participants) | 13 | 12 | 11 | 15 | 14 | 14 | 12 | 14 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 11 | 15 | 14 | 14 | 12 | 14 | 105
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 6 | 9 | 7 | 10 | 6 | 8 | 60
  Male | 6 | 5 | 5 | 6 | 7 | 4 | 6 | 6 | 45

OUTCOME MEASURES:

1. Primary Outcome: Cmax of BIA 9-1067 - Maximum Observed Plasma Concentration of BIA 9-1067 (Day 1)
Description: Cmax - maximum observed plasma concentration following single (Day 1) oral administrations of 5, 25 and 50 mg OPC in healthy Japanese and matched healthy Caucasian subjects Blood samples collected for PK analysis at the following timepoints: on Day 1 at pre-dose (within 1 hour before dose administration) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, and 24 hours post-dose.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Caucasian 5 mg OPC | Caucasian 25 mg OPC | Caucasian 50 mg OPC | Japanese 5 mg OPC | Japanese 25 mg OPC | Japanese 50 mg OPC
Number analyzed (Participants) | 13 | 11 | 11 | 14 | 14 | 12
ng/mL | 182 (64.5) | 794 (392) | 1540 (493) | 176 (93.6) | 797 (323) | 1736 (381)

2. Primary Outcome: Cmax of BIA 9-1067 - Maximum Observed Plasma Concentration of BIA 9-1067 (Day 10)
Description: Cmax - maximum observed plasma concentration following Last (Day 10) oral administrations of 5, 25 and 50 mg OPC in healthy Japanese and matched healthy Caucasian subjects.
  Blood samples collected for PK analysis at the following timepoints: Day 10 at pre-dose (within 1 hour before dose administration) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, and 144 hours post-dose
Time Frame: Day 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Caucasian 5 mg OPC | Caucasian 25 mg OPC | Caucasian 50 mg OPC | Japanese 5 mg OPC | Japanese 25 mg OPC | Japanese 50 mg OPC
Number analyzed (Participants) | 13 | 12 | 11 | 14 | 13 | 12
ng/mL | 226 (110) | 774 (361) | 1550 (655) | 276 (130) | 959 (273) | 1785 (431)

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve (AUC) From Time Zero to Last Time Point With Concentrations Above the Lower Limit of Quantitation of BIA 9-1067 (Day 1)
Description: AUC0-t - area under the concentration-time curve (AUC) from time zero to last time point with concentrations above the lower limit of quantitation of BIA 9-1067 following single (Day 1) oral administrations of 5, 25 and 50 mg OPC in healthy Japanese and matched healthy Caucasian subjects.
  Blood samples collected for PK analysis at the following timepoints: on Day 1 at pre-dose (within 1 hour before dose administration) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, and 24 hours post-dose.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Caucasian 5 mg OPC | Caucasian 25 mg OPC | Caucasian 50 mg OPC | Japanese 5 mg OPC | Japanese 25 mg OPC | Japanese 50 mg OPC
Number analyzed (Participants) | 13 | 11 | 11 | 14 | 14 | 12
ng.h/mL | 267 (113) | 2013 (800) | 3727 (1726) | 319 (154) | 1886 (692) | 4438 (1151)

4. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve (AUC) From Time Zero to Last Time Point With Concentrations Above the Lower Limit of Quantitation of BIA 9-1067 (Day 10)
Description: AUC0-t - Area Under the Concentration-time Curve (AUC) From Time Zero to Last Time Point With Concentrations Above the Lower Limit of Quantitation of BIA 9-1067 following Last (Day 10) oral administrations of 5, 25 and 50 mg OPC in healthy Japanese and matched healthy Caucasian subjects.
  Blood samples collected for PK analysis at the following timepoints: Day 10 at pre-dose (within 1 hour before dose administration) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, and 144 hours post-dose
Time Frame: Day 10
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Caucasian 5 mg OPC | Caucasian 25 mg OPC | Caucasian 50 mg OPC | Japanese 5 mg OPC | Japanese 25 mg OPC | Japanese 50 mg OPC
Number analyzed (Participants) | 13 | 12 | 11 | 14 | 13 | 12
ng.h/mL | 349 (169) | 2024 (820) | 3999 (1770) | 441 (139) | 2222 (407) | 4464 (932)

5. Primary Outcome: AUC0-∞ - Area Under the Concentration of BIA 9-1067-time Curve (AUC) From Time Zero to Infinity (Day 1)
Description: AUC0-∞ - area under the concentration of BIA 9-1067-time curve (AUC) from time zero to infinity following single (Day 1) oral administrations of 5, 25 and 50 mg OPC in healthy Japanese and matched healthy Caucasian subjects Blood samples collected for PK analysis at the following timepoints: on Day 1 at pre-dose (within 1 hour before dose administration) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, and 24 hours post-dose
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Caucasian 5 mg OPC | Caucasian 25 mg OPC | Caucasian 50 mg OPC | Japanese 5 mg OPC | Japanese 25 mg OPC | Japanese 50 mg OPC
Number analyzed (Participants) | 10 | 11 | 11 | 11 | 13 | 12
ng.h/mL | 338 (48.6) | 2039 (798) | 3756 (1734) | 357 (163) | 1976 (673) | 4470 (1147)

6. Primary Outcome: AUC0-∞ - Area Under the Concentration of BIA 9-1067-time Curve (AUC) From Time Zero to Infinity (Day 10)
Description: AUC0-∞ - Area Under the Concentration of BIA 9-1067-time Curve (AUC) From Time Zero to Infinity following Last (Day 10) oral administrations of 5, 25 and 50 mg OPC in healthy Japanese and matched healthy Caucasian subjects.
  Blood samples collected for PK analysis at the following timepoints: Day 10 at pre-dose (within 1 hour before dose administration) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, and 144 hours post-dose
Time Frame: Day 10
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Caucasian 5 mg OPC | Caucasian 25 mg OPC | Caucasian 50 mg OPC | Japanese 5 mg OPC | Japanese 25 mg OPC | Japanese 50 mg OPC
Number analyzed (Participants) | 13 | 12 | 11 | 14 | 13 | 12
ng.h/mL | 409 (147) | 2056 (817) | 4028 (1786) | 465 (145) | 2240 (406) | 4510 (938)

7. Primary Outcome: Tmax of BIA 9-1067 - Time Taken to Reach Maximum Observed Plasma Concentration of BIA 9-1067 (Day 1)
Description: Tmax of BIA 9-1067 - time taken to reach maximum observed plasma concentration following single (Day 1) oral administrations of 5, 25 and 50 mg OPC in healthy Japanese and matched healthy Caucasian subjects.
  Blood samples collected for PK analysis at the following timepoints: on Day 1 at pre-dose (within 1 hour before dose administration) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, and 24 hours post-dose
Time Frame: Day 1
Measure: Median (Full Range); unit: hours
Arm/Group | Caucasian 5 mg OPC | Caucasian 25 mg OPC | Caucasian 50 mg OPC | Japanese 5 mg OPC | Japanese 25 mg OPC | Japanese 50 mg OPC
Number analyzed (Participants) | 13 | 11 | 11 | 14 | 14 | 12
hours | 2.0 [0.75 to 5.0] | 2.0 [1.5 to 4.0] | 3.0 [1.5 to 3.0] | 2.0 [1.0 to 5.0] | 2.0 [1.0 to 8.0] | 2.0 [0.75 to 5.0]

8. Primary Outcome: Tmax of BIA 9-1067 - Time Taken to Reach Maximum Observed Plasma Concentration of BIA 9-1067 (Day 10)
Description: Tmax of BIA 9-1067 - Time Taken to Reach Maximum Observed Plasma Concentration of BIA 9-1067 following Last (Day 10) oral administrations of 5, 25 and 50 mg OPC in healthy Japanese and matched healthy Caucasian subjects.
  Blood samples collected for PK analysis at the following timepoints: Day 10 at pre-dose (within 1 hour before dose administration) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, and 144 hours post-dose
Time Frame: Day 10
Measure: Median (Full Range); unit: hours
Arm/Group | Caucasian 5 mg OPC | Caucasian 25 mg OPC | Caucasian 50 mg OPC | Japanese 5 mg OPC | Japanese 25 mg OPC | Japanese 50 mg OPC
Number analyzed (Participants) | 13 | 12 | 11 | 14 | 13 | 12
hours | 1.00 [0.50 to 5.00] | 2.00 [1.00 to 4.00] | 1.50 [0.50 to 3.00] | 2.00 [0.75 to 5.00] | 2.00 [0.50 to 4.00] | 2.00 [1.00 to 4.00]

ADVERSE EVENTS:
Arm/Group | Caucasian 5 mg OPC | Caucasian 25 mg OPC | Caucasian 50 mg OPC | Caucasian Placebo | Japanese 5 mg OPC | Japanese 25 mg OPC | Japanese 50 mg OPC | Japanese Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/11 | 0/15 | 0/14 | 0/14 | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 7/13 | 5/12 | 6/11 | 8/15 | 3/14 | 6/14 | 6/12 | 5/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Caucasian 5 mg OPC (N=13) | Caucasian 25 mg OPC (N=12) | Caucasian 50 mg OPC (N=11) | Caucasian Placebo (N=15) | Japanese 5 mg OPC (N=14) | Japanese 25 mg OPC (N=14) | Japanese 50 mg OPC (N=12) | Japanese Placebo (N=14)
Vessel puncture site haematoma (General disorders) | 4 | 3 | 0 | 2 | 1 | 2 | 3 | 2
Vessel puncture site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stifness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Eyelid irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Energy increased (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tenderness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laceratioin (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other